CLINICAL TRIAL: NCT06812689
Title: The Acute Effects of Cocoa Flavanols Intake on Overt and Covert Attention: a Randomized, Double-blind Crossover Trial
Brief Title: The Acute Effects of Cocoa Flavanols Intake on Overt and Covert Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Oğuz Karataş, Principal Investigator, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 122K636
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy Young Adults
Keywords: cocoa flavanols; overt attention; covert attention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Baseline/Placebo/Flavanol (Experimental): Participants consumed sugar water, an alkalized cocoa beverage, and a natural cocoa beverage containing 710 mg of flavanols, with a one-week washout period between interventions.
  Interventions: Dietary Supplement: Flavanol; Dietary Supplement: Placebo; Other: Sugar water
- Baseline/Flavanol/Placebo (Experimental): Participants consumed sugar water, a natural cocoa beverage containing 710 mg of flavanols, and an alkalized cocoa beverage, with a one-week washout period between interventions.
  Interventions: Dietary Supplement: Flavanol; Dietary Supplement: Placebo; Other: Sugar water
- Placebo/Baseline/Flavanol (Experimental): Participants consumed an alkalized cocoa beverage, sugar water, and a natural cocoa beverage containing 710 mg of flavanols, with a one-week washout period between interventions.
  Interventions: Dietary Supplement: Flavanol; Dietary Supplement: Placebo; Other: Sugar water
- Placebo/Flavanol/Baseline (Experimental): Participants consumed an alkalized cocoa beverage, a natural cocoa beverage containing 710 mg of flavanols, and sugar water, with a one-week washout period between interventions.
  Interventions: Dietary Supplement: Flavanol; Dietary Supplement: Placebo; Other: Sugar water
- Flavanol/Baseline/Placebo (Experimental): Participants consumed a natural cocoa beverage containing 710 mg of flavanols, sugar water, and an alkalized cocoa beverage, with a one-week washout period between interventions.
  Interventions: Dietary Supplement: Flavanol; Dietary Supplement: Placebo; Other: Sugar water
- Flavanol/Placebo/Baseline (Experimental): Participants consumed a natural cocoa beverage containing 710 mg of flavanols, an alkalized cocoa beverage, and sugar water, with a one-week washout period between interventions.
  Interventions: Dietary Supplement: Flavanol; Dietary Supplement: Placebo; Other: Sugar water

INTERVENTIONS:
Dietary Supplement: Flavanol — Natural cocoa powder containing 710 mg of flavanols was dissolved in 250 mL of hot water and sweetened with 6 g of sugar.
Dietary Supplement: Placebo — Alkalized cocoa powder containing no flavanols was dissolved in 250 mL of hot water and sweetened with 6 g of sugar.
Other: Sugar water — 250 mL of hot water with 6 g of sugar

SUMMARY:
The present study aimed to examine whether a cocoa beverage containing 710 mg of flavanols enhances both overt and covert attention in healthy young adults, using a randomized, double-blind, baseline- and placebo-controlled crossover design.

DETAILED DESCRIPTION:
Cocoa flavanols (CF) have various physiological effects that may directly or indirectly enhance cognitive functions. Following CF intake, a series of biochemical processes within vascular smooth muscle cells lead to the relaxation of smooth muscles, the dilation of blood vessels, and an increase in cerebral blood flow. For the brain to function optimally, cerebral blood flow must be maintained at a level that ensures a constant supply of oxygen and glucose to neurons. During periods of intense neuronal activity, neurons require more oxygen and nutrients, which is met by an increase in blood flow. Given that CF has been shown to enhance blood flow and perfusion in brain regions associated with attention (e.g., the parietal cortex, anterior cingulate cortex, and dorsolateral prefrontal cortex), it was hypothesized that CF intake could acutely improve both overt and covert attention.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal visual acuity

Exclusion Criteria:

* History of neurological, psychiatric, cardiovascular or metabolic disorders
* Following a medically restricted diet
* Taking antidepressant, anxiolytic, and antipsychotic drugs in the past three months
* Currently taking anticoagulant
* Taking herbal supplements in the past week
* Allergic or intolerant to cocoa, caffeine, sucrose, or fructose
* Color blindness

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-26 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Spatial cueing task - accuracy | 1 hour 40 minutes post-ingestion
  Difference in the total accuracy (%)
Spatial cueing task - reaction time | 1 hour 40 minutes post-ingestion
  Difference in the reaction time (ms) for correct responses
Visual search task - accuracy | 1 hour 40 minutes post-ingestion
  Difference in the total accuracy (%)
Visual search task - reaction time | 1 hour 40 minutes post-ingestion
  Difference in the reaction time (ms) for correct responses

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Karataş, Ph.D., Principal Investigator — Konya Necmettin Erbakan University
Locations (1):
- Konya Necmettin Erbakan University Cognitive Psychology Laboratuary, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months after publication with no end date.
Access Criteria: A proposal that describes planned analyses must be submitted

REFERENCES:
- [Background] Karataş O, Karabay A, Alıcı T. Uzun süreli kakao flavanolleri alımının bilişsel işlevlere ve duygudurumuna etkileri ve bu etkilerin altındaki fizyolojik mekanizmalar: Bir derleme çalışması. Türk Psikoloji Yazıları. 2022;25(49):1-26. http://dx.doi.org/10.31828/tpy1301996120211203m000043
- [Background] Lamport DJ, Pal D, Moutsiana C, Field DT, Williams CM, Spencer JP, Butler LT. The effect of flavanol-rich cocoa on cerebral perfusion in healthy older adults during conscious resting state: a placebo controlled, crossover, acute trial. Psychopharmacology (Berl). 2015 Sep;232(17):3227-34. doi: 10.1007/s00213-015-3972-4. Epub 2015 Jun 7. PMID 26047963
- [Background] Francis ST, Head K, Morris PG, Macdonald IA. The effect of flavanol-rich cocoa on the fMRI response to a cognitive task in healthy young people. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S215-20. doi: 10.1097/00005344-200606001-00018. PMID 16794461